CLINICAL TRIAL: NCT02113644
Title: Prevent CardioKids
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Prevent CardioKids
Record Dates: First submitted 2013-10-23; First posted 2014-04-14 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Overweight or obese children: Overweight or obese children according to the International Obesity Task Force (IOTF) criteria following the lifestyle intervention in the Centre for Overweight Adolescent and Children's Healthcare
  Interventions: Other: Lifestyle intervention
- Lean children: Lean children according to the International Obesity Task Force (IOTF) criteria admitted at de pediatric ward for a planned surgery, for example the correction of floppy ears

INTERVENTIONS:
Other: Lifestyle intervention
  Groups: Overweight or obese children

SUMMARY:
The aim of Prevent CardioKids is to evaluate to what extend disturbed vascular function markers are already present in children of different weight categories and whether these are age dependent. Also differences - and relationships - between vascular function measurements and plasma biomarkers between lean and overweight/obese children will be compared.

DETAILED DESCRIPTION:
The aim of Prevent CardioKids is to evaluate to what extend disturbed vascular function markers are already present in children of different weight categories and whether these are age dependent. Also differences - and relationships - between vascular function measurements and plasma biomarkers between lean and overweight/obese children will be compared.The primary endpoint is to examine the difference in micro- and macro-vasculature characteristics in children with different weight classifications (lean; overweight; obese; extreme obese; morbid obese). Secondary endpoints are differences in lipoprotein profiles, pro-inflammatory and oral glucose tolerance profiles between different age groups, between lean and overweight/obese children and in relation with the measured micro- and macro-vasculature characteristics

ELIGIBILITY:
Inclusion Criteria:

* Participation in the COACH program
* Aged between 6 and 18 years (at time of inclusion)
* Overweight or obesity according to IOTF criteria

In order to be eligible to participate in the control group, a subject must meet all of the following criteria:

* Aged between 6 and 18 years
* Normal weight according to the IOTF criteria
* Undergo surgery for elective reasons

Exclusion Criteria:

* Retarded children
* Children suffering from:

  * Inflammatory diseases: auto-immune diseases, inflammatory bowel diseases, hepatitis, dermatitis, nephritis, pancreatitis, gastro-enteritis, vasculitis, salpingitis, arthritis, osteomyelitis, myositis, ear-nose-throat infections
  * Allergic diseases: asthma, eczema, hay fever, food allergies
  * Oncologic diseases
  * Cystic fibrosis
  * Type 1 diabetes mellitus
  * Congenital metabolic diseases
* Malnourished children

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Overweight or obese children according to the International Obesity Task Force (IOTF) criteria between 6-18 years old. Overweight and obese children will be recruited in the COACH program. For the control group healthy, normal weight children between 6-18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2014-04; Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Vascular function measured by peripheral arterial tonometry (EndoPAT) | 1 year
  The primary endpoint is the difference in micro- and macrovascular characteristics, as measured by EndoPAT in lean/overweight/obese children in different age groups.

SECONDARY OUTCOMES:
Differences in characteristics of the microcirculation as measured via fundus photography | 1 year
  Differences in characteristics of the microcirculation as measured via fundus photography in overweight/obese children in different age groups, between lean and overweight/obese children in different age groups and in relation with the measured micro- and macrovascular characteristics
Differences in characteristics of microcirculation measured via lipoprotein profiles | 1 year
  Differences in characteristics of the microcirculation as measured via lipoprotein profiles in overweight/obese children in different age groups, between lean and overweight/obese children in different age groups and in relation with the measured micro- and macrovascular characteristics
Differences in characteristics of the microcirculation as measured via pro-inflammatory profiles | 1 year
  Differences in characteristics of the microcirculation as measured via pro-inflammatory profiles in overweight/obese children in different age groups, between lean and overweight/obese children in different age groups and in relation with the measured micro- and macrovascular characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Anita Vreugdenhil, dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- See also: Related Info — http://www.coachmaastricht.com